CLINICAL TRIAL: NCT04482777
Title: IL37,Tlymphocytes ,NK Cells in Pathogenesis of Immune Thrombocytopenia.
Brief Title: IL37,Tlymphocytes,NK Cells in Pathogenesis of ITP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Mohamed Elsayed, Resident physician, Assiut University
Other Study IDs: Cellular immunity in ITP
Record Dates: First submitted 2020-07-19; First posted 2020-07-23 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: ITP

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ITP: Patient newly diagnosied with ITP
  Interventions: Drug: Corticosteriod for treated patients
- Treated: Patients with ITP recived treatment
  Interventions: Drug: Corticosteriod for treated patients
- Control: Healthy people
  Interventions: Drug: Corticosteriod for treated patients

INTERVENTIONS:
Drug: Corticosteriod for treated patients — Drug given to some patients with autoimmune disease

SUMMARY:
To evaluate the role of IL37 in pathogenesis of ITP and to study the relation between IL37,Tlymphocytes,NK cells in ITP

DETAILED DESCRIPTION:
Idiopathic thrombocytopenia or immune thrombocytopenia (ITP) is a hematological condition which is characterized by a low platelet count of less than 100 x 109L . Symptoms of ITP can vary but tend to be symptoms of thrombocytopenia in general, such as petechiae, purpura, mucosal bleeding and in the most severe cases fatal intracranial hemorrhage(1,2) Interleukin (IL)-37, a novel anti-inflammatory cytokine previously known as interleukin-1 family member 7 before it was renamed, has a pivotal role in the suppression of immune responses (3,4). IL-37 is widely expressed in several types of cells, tissues and organs, including peripheral blood mononuclear cells (PBMCs) (5). The major role of IL-37 is to decrease excessive inflammation in innate and adaptive immune diseases, mainly by inhibiting the expression, production and function of pro-inflammatory cytokines, including IL-1α, IL-6, tumor necrosis factor (TNF) and macrophage inflammatory protein-2. The abundance of these cytokines has been reported to increase with the silencing of endogenous IL-37 in human blood cells (3,6).Aberrant expression of IL-37 has been observed in several inflammatory and autoimmune diseases However, the role of IL-37 in ITP has remained elusive. Immune thrombocytopenia pathogenesis is a complicated process. T cell immune abnormalities are involved in ITP pathogenesis. These abnormalities include platelet auto-antigen reactive cytotoxic T cells, abnormal numbers and functions of T regulatory cells, loss of Th1/Th2 balance, megakaryocyte maturation abnormalities and abnormal T cell anergy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ITP (moderate and sever) different age group.

Exclusion Criteria:

* Patients with stroke and myocardial infarction,malignant tumors or pregnancy.

Ages: 2 Years to 60 Years | Sex: All
Age Groups: Child, Adult
Study Population: To study initially enrolled 90 patients with ITP in Assiut hospital
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-07-30 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
To decrease the immunity complications in ITP patients | Baseline
  Early detection of immunity complications in ITP patients
To decrease case fatality rate | Baseline
  Early detection of immunity complication will decrease mortality rate

REFERENCES:
- [Background] Lambert MP, Gernsheimer TB. Clinical updates in adult immune thrombocytopenia. Blood. 2017 May 25;129(21):2829-2835. doi: 10.1182/blood-2017-03-754119. Epub 2017 Apr 17. PMID 28416506
- [Background] Kistangari G, McCrae KR. Immune thrombocytopenia. Hematol Oncol Clin North Am. 2013 Jun;27(3):495-520. doi: 10.1016/j.hoc.2013.03.001. PMID 23714309
- [Background] Chen Z, Qu W, Wang HQ, Xing LM, Wu YH, Liu ZY, Zhang Y, Liu H, Dong XF, Tao JL, Shao ZH. [Relationship of Peripheral Blood IL-37 Expression with T Lymphocytes Subsets and NK Cells in Patients with Primary Immune Thrombocytopenia]. Zhongguo Shi Yan Xue Ye Xue Za Zhi. 2019 Aug;27(4):1201-1207. doi: 10.19746/j.cnki.issn.1009-2137.2019.04.034. Chinese. PMID 31418380
- [Background] Zhao Y, Ni X, Xu P, Liu Q, Sun T, Liu X, Ji X, Qiu J, Li J, Wang S, Han P, Peng J, Hou M, Li G. Interleukin-37 reduces inflammation and impairs phagocytosis of platelets in immune thrombocytopenia (ITP). Cytokine. 2020 Jan;125:154853. doi: 10.1016/j.cyto.2019.154853. Epub 2019 Sep 23. PMID 31557634